CLINICAL TRIAL: NCT05497063
Title: Randomized, Single Oral Dose, Open-label, Single-period, Parallel Group, Bioequivalence Study to Compare Sulfadoxine/Pyrimethamine Two Dispersible Tablets (250 mg Sulfadoxine / 12.5 mg Pyrimethamine) Versus G-COSPE® One Tablet (500 mg Sulfadoxine / 25 mg Pyrimethamine) in Healthy Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Sulfadoxine/ Pyrimethamine Dispersible Tablets in Healthy Subjects Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Emzor Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1100-2021
Record Dates: First submitted 2022-05-01; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Sulfadoxine; Pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulfadoxine/Pyrimethamine dispersible tablets, 250 mg sulfadoxine / 12.5 mg pyrimethamine (Experimental): Two dispersible tablets of Sulfadoxine/Pyrimethamine (250 mg sulfadoxine / 12.5 mg pyrimethamine to be given as single dose once under fasting condition
  Interventions: Drug: Sulfadoxine/Pyrimethamine dispersible tablets, 250 mg sulfadoxine / 12.5 mg pyrimethamine & 500 mg sulfadoxine / 25 mg pyrimethamine
- G-COSPE® tablets, 500 mg sulfadoxine / 25 mg pyrimethamine (Active Comparator): One tablet of G-COSPE® tablets, 500 mg sulfadoxine / 25 mg pyrimethamine to be given as single dose once under fasting condition
  Interventions: Drug: G-COSPE® tablets

INTERVENTIONS:
Drug: Sulfadoxine/Pyrimethamine dispersible tablets, 250 mg sulfadoxine / 12.5 mg pyrimethamine & 500 mg sulfadoxine / 25 mg pyrimethamine — Two tablets of 250 mg sulfadoxine / 12.5 mg pyrimethamine or 500 mg sulfadoxine / 25 mg pyrimethamine to be given as single dose once under fasting condition
  Arms: Sulfadoxine/Pyrimethamine dispersible tablets, 250 mg sulfadoxine / 12.5 mg pyrimethamine
Drug: G-COSPE® tablets — One tablet of G-COSPE® tablets, 500 mg sulfadoxine / 25 mg pyrimethamine to be given as single dose once under fasting condition
  Arms: G-COSPE® tablets, 500 mg sulfadoxine / 25 mg pyrimethamine

SUMMARY:
To asses bio equivalence between two (500 mg sulfadoxine / 25 mg pyrimethamine) formulation

DETAILED DESCRIPTION:
• The aim of this study is to assess bioequivalence between a single dose from the test product, Sulfadoxine/Pyrimethamine two dispersible tablets (250 mg sulfadoxine / 12.5 mg pyrimethamine), manufactured by Emzor Pharmaceuticals Industries Ltd, Nigeria versus the reference product G-COSPE® one tablet (500 mg sulfadoxine / 25 mg pyrimethamine) manufactured by Guilin Pharmaceutical Co. Ltd, China.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject is Caucasian & aged between eighteen & fifty years (18 - 50), both inclusive.

  2. The subject is within the limits for his/her height & weight as defined by the body mass index range (18.5 - 30.0 Kg/m2).

  3. The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.

  4. Results of medical history, vital signs, physical examination & conducted medical laboratory tests are normal as per appendix 3.

  5. The subject tested negative for hepatitis (B & C) viruses and human immunodeficiency virus (HIV).

  6. There is no history or evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.

  7. The subject is able to understand and willing to sign the informed consent form.

  8. The subject has normal liver (AST & ALT enzymes) function. 9. The subject's kidney function tests are within normal ranges. As per appendix 3.

  10. The subject has normal respiratory system. 11. The subject's folic acid levels are within normal range. 12. The subject has normal platelet levels. As per appendix 3. 13. For female subjects: negative pregnancy test and the woman is using two reliable contraception methods during the study and until 52 days after dosing.

Note: Pyrimethamine/sulfadoxine showed reproductive toxicity in animal studies. Pyrimethamine/sulfadoxine should not be used during the first trimester of pregnancy unless the benefit is considered to outweigh the risks and alternative drugs are not available. During 2nd or 3rd trimesters of pregnancy, may be used for intermittent preventive treatment in pregnancy.

14. The subject has normal cardiovascular system, ECG recording & QTc interval less than 450 ms.

Exclusion Criteria:

* 1. The subject is a heavy smoker (more than 10 cigarettes per day). 2. The subject has suffered an acute illness one week before dosing. 3. The subject has a history of or concurrent consumption of alcohol. 4. The subject has a history of or concurrent consumption of illicit drugs. 5. The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.

  6. Subject who has been hospitalized within three months before the study or during the study.

  7. Subject who is vegetarian. 8. The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 72 hours after dosing.

  9. The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing and any time during the study, unless otherwise judged acceptable by the clinical investigator.

  10. The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before dosing and any time during the study.

  11. The subjects who have been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study 12. The subjects who have donated blood within 80 days before first dosing. 13. The subject has a history of G6PD Deficiency. 14. The subject has a history presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Peak Plasma Concentration (Cmax) for Sulfadoxine and Pyrimethamine. | 72 hours
  The average bioequivalence of the products will be concluded if the two-sided 90 % confidence interval for the test to reference ratio of the population means is within 80.00 - 125.00 % for the ln transformed data Cmax of sulfadoxine & pyrimethamine
Area under the plasma concentration versus time curves (AUC0 - 72) for Sulfadoxine and Pyrimethamine | 72 hours
  The average bioequivalence of the products will be concluded if the two-sided 90 % confidence interval for the test to reference ratio of the population means is within 80.00 - 125.00 % for the ln transformed data AUC0 -72 of sulfadoxine & pyrimethamine

SECONDARY OUTCOMES:
Obtaining the Tmax (Time to reach maximum concentration) for Sulfadoxine and Pyrimethamine | 72 hours
  The descriptive statistics including Maximum, Minimum and Median values will be measured for Tmax
Number of participant with treatment related adverse events as assessed by CTCAE v4.0. | ECG recording will be performed 4 hours post- dosing and at the end of the study (at 72.00 hours post dosing) as follow-up tests
  ECG QTc Interval (safety and tolerability) Clinically significant abnormal deviations in ECG QTc interval
Number of participant with treatment related adverse events as assessed by CTCAE v4.0. | At 1-hour pre-dosing; 2, 4, 6, 8, 12 and 23 hours post-dosing (±45 minutes of scheduled time). Blood pressure will also be measured at 48 and 72 hours post-dosing upon ambulatory sample collection.
  Blood pressure (safety and tolerability) Clinically significant abnormal deviations. Normal range of blood pressure > 90/60 and <140/90 mmHg. Treatment will be offered to those subjects whom blood pressure drops to 90/60 mm Hg or less and the subject will be excluded in case of not responding to treatment
Number of participant with treatment related adverse events as assessed by CTCAE v4.0. | At 1-hour pre-dosing; 2, 4, 6, 8, 12 and 23 hours post-dosing (±45 minutes of scheduled time). Pulse will also be measured at 48 and 72 hours post-dosing upon ambulatory sample collection.
  Pulse (safety and tolerability) Clinically significant abnormal deviations. Normal range of Pulse 60-100 Bpm
Number of participant with treatment related adverse events as assessed by CTCAE v4.0. | At 1-hour pre-dosing; 2, 6, 10, 14, 18, 22 & 23 hours postdosing (±45 minutes of scheduled time).Temperature will also be measured at 48 and 72 hours post-dosing upon ambulatory sample.
  Temperature (safety and tolerability) Clinically significant abnormal deviations. The temperature will be measured axillary, orally or using infrared thermometer, standardized across all subjects. Normal range of temperature 36.5-37.5 ºC.
Number of participant with treatment related adverse events as assessed by CTCAE v4.0. | At 1-hour pre-dosing; 2, 6, 10, 14, 18, 22 & 23 hours postdosing (±45 minutes of scheduled time).Respiratory rate will also be measured at 48 and 72 hours post-dosing upon ambulatory sample.
  Respiratory rate (safety and tolerability) Clinically significant abnormal deviations. Normal range of respiratory rate 12-18 B/M
Number of participant with treatment related adverse events as assessed by CTCAE v4.0. | At the end of the study (at 72.00 hours post dosing
  Hematology (Safety and Tolerability) Hematology test will include Complete blood count

IPD SHARING:
Plan to Share IPD: No